CLINICAL TRIAL: NCT02691377
Title: Efficacy and Safety of Acupuncture for Primary Sjögren Syndrome
Brief Title: Acupuncture for Primary Sjögren Syndrome
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Responsible Party: Principal Investigator, Zhou Xinyao, Attending Physician & Lecturer, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2015S320
Record Dates: First submitted 2016-02-20; First posted 2016-02-25 (Estimated); Last update posted 2016-02-29 (Estimated); Status verified 2016-02

CONDITIONS: Sjogren's Syndrome
MeSH Terms: conditions — Sjogren's Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acupuncture group (Experimental): Participants will receive acupuncture for 8 weeks. In particular, acupuncture will be performed three times a week in earlier 4 weeks and twice a week in later 4 weeks.
  Interventions: Device: acupuncture group
- Sham Acupuncture group (Sham Comparator): Participants will receive sham acupuncture for 8 weeks. The procedure is the same as the acupuncture arm.
  Interventions: Device: Sham Acupuncture group

INTERVENTIONS:
Device: acupuncture group — Acupoints include 11 on the head, two on the upper extremities, and two on the lower extremities. Before performing acupuncture, a small pad will be pasted on each acupoint. All the needles will insert the acupoints through these pads. Then, they will be twirled, lifted and thrust three times to elicit the Deqi sensation. Each session will last 30 minutes.
  Arms: Acupuncture group
Device: Sham Acupuncture group — The same acupoints with acupuncture group are selected.A placebo needle with a blunt tip will be used to perform sham acupuncture. They will only insert the pad and no skin penetration. The same procedure with acupuncture group will be performed.
  Arms: Sham Acupuncture group

SUMMARY:
The purpose of this study is to determine whether acupuncture is effective and safe in the treatment of Primary Sjögren Syndrome.

DETAILED DESCRIPTION:
This randomized, double-blinded, sham acupuncture controlled trial is aimed to assess the effectiveness and safety of acupuncture in the treatment of Primary Sjögren Syndrome.The eligible participants will be randomly allocated to receive acupuncture or sham acupuncture for 8 weeks.

Assuming a two-sided alpha of 0.05, power of 85%, and a 20% drop-out, a sample sized of 30 would be needed for each group. The statistical analysis will be based on the intention-to-treat principle. Continuous variables will be compared by Student t test or Mann-Whitney U test; categorical variables will be analyzed by chi-square test, Fisher's exact test or Kruskal-Wallis H test as appropriate. For comparison between two time points, paired t-test or Wilcoxon signed rank test will be used as appropriate. A statistically significant difference was set at P<0.05.

ELIGIBILITY:
Inclusion Criteria:

* To fulfill the American-European Consensus Group Criteria for primary Sjögren syndrome.
* With the symptoms of primary Sjögren syndrome less than 5 years.

Exclusion Criteria:

* With an acupuncture contraindication (allergy to metals, skin lesions on relative acupoints, etc.)
* Taking or taken medicine for primary Sjögren syndrome within last 4 weeks before the enrollment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-03; Primary Completion 2017-03 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
The proportion of participants who has a 30% or greater reduction in 2 of 3 items,including the numeric analog scale (NAS) of dryness, fatigue, and pain. | 24 weeks
  Subjects will be asked to provide every NAS score based on the average situation over the past 24 hours 13 rather than a point of time. And we will collect NAS scores three times a week in week0-8 (24 times in total) as removal of a variety of factors causing bias, including mental relaxation in weekend, weather changing, or unexpected events life in, etc., each of which may influence the feelings of dryness, fatigue, and pain.

SECONDARY OUTCOMES:
Change in NAS of each item including dryness, fatigue, and pain. | 24 weeks
  Subjects will be asked to provide every NAS score based on the average situation over the past 24 hours 13 rather than a point of time. And we will collect NAS scores three times a week in week0-8 (24 times in total) as removal of a variety of factors causing bias, including mental relaxation in weekend, weather changing, or unexpected events life in, etc., each of which may influence the feelings of dryness, fatigue, and pain.
Change in EULAR Sjögren's Syndrome Patient Reported Index (ESSPRI) | 24 weeks
  it will be measured at week0/8/16/24
Change in Medical Outcome Study Short Form 36 Short-Form Health Survey (SF-36) | 24 weeks
  it will be measured at week0/8/16/24
Change in Hospital Anxiety and Depression (HAD) scale score | 24 weeks
  it will be measured at week0/8/16/24
Change in serum Immunoglobulin G (IgG),immunoglobulin A (IgA), and immunoglobulin M (IgM) levels | 24 weeks
  it will be measured at week0/24
Change in image of Salivary glands measured by ultrasound | 24 weeks
  it will be measured at week0/24
Change in Schirmer test score and unstimulated salivary flow | 24 weeks
  it will be measured at week0/8/16/24
Adverse events | 24 weeks
  it will be measured at week0/8/16/24, and be observed, documented, and evaluated in detail.

CONTACTS AND LOCATIONS:
Overall Officials: Xinyao Zhou, MD, Principal Investigator — Guang'anmen Hospital
Locations (1):
- Guang'anmen Hospital, China academy of Chinese Medical Sciences, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zhou X, Xu H, Chen J, Wu H, Zhang Y, Tian F, Tang X, Zhang H, Ge L, Li K, Jiang W, Liu Z, Jiang Q. Efficacy and Safety of Acupuncture on Symptomatic Improvement in Primary Sjogren's Syndrome: A Randomized Controlled Trial. Front Med (Lausanne). 2022 May 6;9:878218. doi: 10.3389/fmed.2022.878218. eCollection 2022. PMID 35602489
- [Derived] Jiang Q, Zhang H, Pang R, Chen J, Liu Z, Zhou X. Acupuncture for Primary Sjogren Syndrome (pSS) on symptomatic improvements: study protocol for a randomized controlled trial. BMC Complement Altern Med. 2017 Jan 19;17(1):61. doi: 10.1186/s12906-017-1559-9. PMID 28103850